CLINICAL TRIAL: NCT05475847
Title: A Phase I Clinical Study to Evaluate Safety and Efficacy of C-TIL052A Cell Therapy (Autologous Tumor Infiltrating Lymphocytes Injection Combined With IL-2) in Subjects With Persistent, Recurrent and/or Metastatic Cervical Cancer
Brief Title: Study of C-TIL052A Cell Therapy in Advanced Cervical Cancer
Acronym: TIL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaohua Wu MD, Professer, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1031-031
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cervical Cancer
Keywords: Gynecological tumor; Tumor Infiltrating Lymphocytes
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-TIL052A treatment group (Experimental): C-TIL052A autologous infiltrating lymphocytes injection followed by injection of Interleukin 2 (IL-2)
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocytes (C-TIL052A) Injection

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocytes (C-TIL052A) Injection — C-TIL052A injection followed by injection of IL-2

SUMMARY:
A study that aimed to assess the safety and anti-tumor activity of C-TIL052A cell therapy in subjects with persistent, recurrent and/or metastatic cervical cancer.

DETAILED DESCRIPTION:
For patients with advanced cervical cancer who have failed the standard treatment, no recognized alternative follow-up treatment regimens are available and the prognosis is poor. The study is a single center phase I trial planning to assess the safety, tolerability and the preliminary anti-tumor activity of C-TIL052A cell therapy in persistent, recurrent and/or metastatic cervical cancer. Eligible subjects will receive injection of C-TIL052A (Autologous Tumor Infiltrating Lymphocytes, TIL) and interleukin 2 (IL-2) after lymphodepletion. All subjects will be followed up post treatment for safety and efficacy monitoring and the follow-up period will be 12 months or through study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years at screening
2. Voluntary participation and able to sign the informed consent form
3. Patients with histologically confirmed persistent, recurrent and/or metastatic cervical cancer who failed the standard treatment.
4. Has access to tumor tissue and can isolate ≥1.0g of tumor tissue mass for the preparation of autologous tumor infiltrating lymphocytes
5. At least one measurable target lesion (per RECIST v1.1)
6. ECOG performance status score: 0~1
7. Expected survival ≥ 3 months
8. Negative serum or urine pregnancy test results for females of child-bearing age at screening

Exclusion Criteria:

1. Uncontrolled CNS disease, severe cerebrovascular disease or obvious neurological symptoms (including mental disease)
2. Symptomic chronic obstructive pulmonary disease or persistent asthma
3. Uncontrolled cardiovascular diseases
4. History of primary immune deficiency, autoimmune disease or chronic inflammatory disease
5. High-risk subjects with rapid tumor progression as judged by the Investigator(s)
6. Complicated with infectious diseases, such as hepatitis B/C, syphilis, AIDS
7. History of organ transplantation or allogeneic cell therapy
8. Any situation judged by the Investigator(s) that will have safety concern or interfere with the study results

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | up to 12 months or through study completion
  To characterize the safety profile and evaluate tolerability of C-TIL052A cell therapy by collecting, analyzing the treatment emergent adverse events (TEAEs) and adverse events of special interest (AESIs) during and post treatment, especially the incidence and severity of adverse events (AE) within 28 days post TIL infusion.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months or through study completion
  Proportion of patients with response (CR+PR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease Control Rate (DCR) | up to 12 months or through study completion
  Proportion of patients ever comfirmed with response or stable disease (CR+PR+SD) during the follow-up period per RECIST v1.1
Duration of Response (DOR) | up to 12 months or through study completion
  The time length between the first confirmed objective response to the treatment and the subsequent disease progression per RECIST 1.1
Time to Response (TTR) | up to 12 months or through study completion
  The time length between TIL infusion and confirmed subsequent disease progression per RECIST 1.1
Overall Survival（OS） | up to 12 months or through study completion
  The time length of patients living from the date of TIL infusion
Progression Free Survival（PFS） | up to 12 months or through study completion
  The time length of patients living without progression from the date of TIL infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, MD, Ph.D, Principal Investigator — Fudan University; Jian Zhang, MD, Ph.D, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, No. 270, Dong'an Road, Xuhui District, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, No. 4333, Kangxin Road, Pudong New Area, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No